CLINICAL TRIAL: NCT03168750
Title: Prospective, Multicenter Study to Assess Performance of a Tapered Porous Coated Stem and a Cementless Hemispherical Acetabular Component in Total Hip Arthroplasty
Brief Title: Analysis of a Tapered Porous Coated Stem and a Cementless Hemispherical Acetabular Component
Status: Completed | Type: Observational
Sponsor: Medacta USA (Industry)
Responsible Party: Sponsor
Other Study IDs: MUSA-H-ML-001
Record Dates: First submitted 2017-05-17; First posted 2017-05-30 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Femoral Component:Medacta Masterloc Stem and Medacta MPACT cup: All patients enrolled will receive the Medacta Masterloc Stem and MPACT cup with Highcross PE liner.
  Interventions: Device: Femoral Component:Medacta Masterloc Stem and Medacta MPACT cup.

INTERVENTIONS:
Device: Femoral Component:Medacta Masterloc Stem and Medacta MPACT cup. — Total hip arthroplasty (THA) is one of the most commonly performed and successful orthopaedic operations in improving a patient's quality of life. Orthopaedic surgeons are continually striving to improve all aspects of care relating to this procedure whether this is improvements in implant technology, instrument improvement, or the technique involved in performing the procedure.The results of this study will establish the performance of the femoral component and acetabular component, and provide a general estimate of survivorship, clinical effectiveness and complications.

SUMMARY:
This prospective study will evaluate the hip function and quality of life of patients operated for total hip arthroplasty with Masterloc femoral stem and MPACT acetabular cup. The results of this study will establish the performance of Masterloc femoral component (Medacta International SA) and MPACT acetabular component (Medacta International SA), and provide a general estimate of survivorship, clinical effectiveness and complications.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of the hip necessitating primary hip replacement,
* Suitability for straight cementless stem,
* Adult male and female under 75 years old,
* Ability to give informed consent ,
* Patients who understand the conditions of the study and are willing to participate for the length of the prescribed follow-up.

Exclusion Criteria:

* Off-label use of the Medacta Masterloc femoral component and MPACT acetabular component
* Post-traumatic deformity in the affected hip,
* Patient suffering from Inflammatory arthritis including rheumatoid arthritis,
* Patient suffering by congenital or developmental deformity,
* Severe osteoporosis,
* History of surgery in the affected hip,
* Perioperative fracture,
* Personality disorders (dementia, alcohol or drug abuse etc) suspected of making completion of the trial uncertain,
* Patients with a history of active infection
* Pregnant women or those seeking to become pregnant

Max Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing surgery as part of routine care.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score (HHS) | pre-operative, 4-8 weeks post-operative, 4-8 months post-operative, 9-15 months post operative, 18-30 months post-operative, 4-6 years post-operative, 9-11 years post-operative.
  Assessment of the improvement of clinical outcomes following total hip replacement using the Harris Hip Score
Hip Disability and Osteoarthritis Outcome Score (HOOS) | pre-operative, 4-8 weeks post-operative, 4-8 months post-operative, 9-15 months post operative, 18-30 months post-operative, 4-6 years post-operative, 9-11 years post-operative.
  Assessment of the improvement in activity levels following total hip replacement using the Hip Disability and Osteoarthritis Outcome Score
Oxford Hip Score (OHS) | pre-operative, 4-8 weeks post-operative, 4-8 months post-operative, 9-15 months post operative, 18-30 months post-operative, 4-6 years post-operative, 9-11 years post-operative.
  Assessment of the improvement in the patients physical level of activity using the Oxford Hip Score
Veterans Rand 12 (VR-12) | pre-operative, 4-8 weeks post-operative, 4-8 months post-operative, 9-15 months post operative, 18-30 months post-operative, 4-6 years post-operative, 9-11 years post-operative.
  Assessment of the improvement in your health using the Veterans Rand 12
EuroQol 5 dimension (EQ-5D) | pre-operative, 4-8 weeks post-operative, 4-8 months post-operative, 9-15 months post operative, 18-30 months post-operative, 4-6 years post-operative, 9-11 years post-operative.
  Assessment of the improvement in quality of life and joint movement using the EQ-5D

SECONDARY OUTCOMES:
Radiographic analysis | pre-operative, 4-8 weeks post-operative, 4-8 months post-operative, 9-15 months post operative, 18-30 months post-operative, 4-6 years post-operative, 9-11 years post-operative.
  Radiographic analysis will include evaluation of osteolysis, radiolucent lines, bone hypertrophy, component migration, heterotopic ossification, resorption of calcar.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Tucson Othropedic Institute, Oro Valley, Arizona
  - Jordan Valley Medical Center of Orthopedics Rehabilitation and Excellence, West Jordan, Utah
  - Spokane Joint Replacement Center, Spokane, Washington